CLINICAL TRIAL: NCT01770496
Title: Age-Specific Strategies for Immunization Reminders and Recalls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kevin Dombkowski, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: U01IP000088-01 (NIH)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Childhood Vaccination
Keywords: immunization; vaccination; immunization information system; immunization registry; reminder / recall

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No reminder / recall notice (No Intervention): No childhood vaccination reminder / recall notification sent. Stratified by age cohort of subjects: 7 month recall; 12 month reminder; 19 month recall
- mailed reminder / recall notice (Experimental): Childhood vaccination reminder / recall notification sent by postal mail. Stratified by age cohort of subjects: 7 month recall; 12 month reminder; 19 month recall
  Interventions: Behavioral: Childhood vaccination reminder / recall notification

INTERVENTIONS:
Behavioral: Childhood vaccination reminder / recall notification
  Other Names: Reminder / recall notifications sent by postal mail
  Arms: mailed reminder / recall notice

SUMMARY:
The objective of this study was to assess the relative effectiveness of reminder/recall strategies among children who live in an urban area targeting alternative age-specific milestones.

ELIGIBILITY:
Inclusion Criteria:

* 7 and 19 month recall groups: children not up to date for at least one vaccination at the time of notification
* 12 month reminder group: 12 months of age at time of notification
* Hib vaccination series was not assessed due to a vaccine shortage

Exclusion Criteria:

* Children were ineligible for notifications if they were designated in the Michigan Care Improvement Registry (MCIR)as having died, documented previously as having moved out of the jurisdiction ("Moved or Gone Elsewhere" (MOGE)), opted out of MCIR by their parent, or if they had been previously mailed for MCIR reminder/recall activity in the prior 60 days.

Ages: 7 Months to 19 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10175 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
new immunization doses | within 60 days of reminder notification
  Receipt of 1 or more childhood vaccinations with administration date following reminder notification date

SECONDARY OUTCOMES:
Cost of vaccination reminder | During the time of reminder notification preparation and mailing and approximately 1 month following mailing
  Estimated personnel costs to generate reminder notifications, print, fold / stuff envelopes and follow up on undeliverable notifications
historical immunization doses | within 60 days of reminder notification
  One or more vaccination recorded with the date of administration prior to the reminder notification date
waived doses | within 60 days of reminder notification
  One or more immunization waiver (non-administration) recorded with the date following the date of reminder notification

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Dombkowski, DrPH, MS, Principal Investigator — University of Michigan, Child Health Evaluation and Research (CHEAR) Unit
Locations (1):
- University of Michigan, Child Health Evaluation and Research (CHEAR) Unit, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Dombkowski KJ, Costello LE, Harrington LB, Dong S, Kolasa M, Clark SJ. Age-specific strategies for immunization reminders and recalls: a registry-based randomized trial. Am J Prev Med. 2014 Jul;47(1):1-8. doi: 10.1016/j.amepre.2014.02.009. Epub 2014 Apr 18. PMID 24750973